CLINICAL TRIAL: NCT02328079
Title: Antiviral Treatment in Facial Palsy. Randomized Control Trial
Brief Title: Steroid-Antiviral Treatment in Rehabilitation of Facial Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Antiviral in facial palsy
Record Dates: First submitted 2014-12-10; First posted 2014-12-31 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Facial Palsy
Keywords: Facial Palsy (acute), Acyclovir, Prednisolone
MeSH Terms: conditions — Facial Paralysis | interventions — Steroids; Prednisolone; Antiviral Agents; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid Group (Active Comparator): prednisolone 60 mg /day IM /IV for 6 consecutive days then reduced by 10 mg /day (for a total treatment time for 12 days)
  Interventions: Drug: Steroids (Prednisolone) and Steroids plus Antiviral (Prednisolone + acyclovir)
- Steroid + Antiviral Group (Active Comparator): Prednisolone IM/ IV 60 mg /day + IV acyclovir 500 mg three time /day for 6 consecutive days) then reduced by 10 mg /day (for a total treatment time for 12 days)
  Interventions: Drug: Steroids (Prednisolone) and Steroids plus Antiviral (Prednisolone + acyclovir)

INTERVENTIONS:
Drug: Steroids (Prednisolone) and Steroids plus Antiviral (Prednisolone + acyclovir) — Group allocations: Steroid group (prednisolone 60 mg /day IM /IV), Steroid plus Antiviral group (Prednisolone IM/ IV 60 mg /day + IV acyclovir 500 mg three time /day for 6 consecutive days) then reduced by 10 mg /day (for a total treatment time for 12 days) were placed in serially-numbered opaque closed envelopes. Each patient was placed in the appropriate group after opening the corresponding sealed envelope.
  Other Names: Steroid group (Prednisolone), Steroid plus Antiviral group (Prednisolone + acyclovir)

SUMMARY:
The purpose of this study is to assess the efficacy of antiviral medicine (acyclovir) in recovery of complete facial Palsy. Fifty patients (Males and females) with acute Facial Palsy within the first 3 days of onset with age ranged from 15-60 years old. Each patient was submitted to the following clinical evaluation using House and Brackmann 6 facial function scoring system and Synnybrook grading system. Neurophysiological assessment of facial nerve and muscles was done before and after the end of treatment, then after the end of first and second month of treatment. EMG was done for facial muscles of both sides beside measuring facial nerve excitability to determine the excitation threshold by recording the minimum electrical stimulus required to produce visible muscle contraction. A difference greater than 3.5 mA between the affected and unaffected side is considered significant in terms of poor prognosis. Nerve conduction study of facial nerves of both sides using concentric needle electrode. Trigeminal Blink reflex for both sides of the face. Facial functional recovery was defined as "good" or "complete" using the same criteria used in the 2001 practice guideline. An outcome of grade I or II was considered a good recovery using the House and Brackmann 6 facial function scoring system

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of antiviral medicine (acyclovir) in recovery of complete facial Palsy. Fifty patients (Males and females) with acute Facial Palsy within the first 3 days of onset with age ranged from 15-60 years old. Each patient was submitted to the following clinical evaluation using House and Brackmann 6 facial function scoring system and Synnybrook grading system. Neurophysiological assessment of facial nerve and muscle was done before and after the end of treatment, then after the end of first and second month of treatment. EMG was done for facial muscles of both sides beside measuring facial nerve excitability to determine the excitation threshold by recording the minimum electrical stimulus required to produce visible muscle contraction. A difference greater than 3.5 mA between the affected and unaffected side is considered significant in terms of poor prognosis. Nerve conduction study of facial nerves of both sides using concentric needle electrode. Trigeminal Blink reflex for both sides of the face. Facial functional recovery was defined as "good" or "complete" using the same criteria used in the 2001 practice guideline. An outcome of grade I or II was considered a good recovery using the House and Brackmann 6 facial function scoring system

ELIGIBILITY:
Inclusion Criteria:

* Acute onset facial palsy within the first three days of onset. Age ranged from 15-60 years old

Exclusion Criteria:

* Patients with brittle diabetes mellitus, Morbid obesity, renal or liver impairment, osteopenia, prior history of steroid intolerance.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Facial muscle function using clinical scale | 2 months
  Evaluations of facial muscle function using clinical scale were performed blindly by a neurologist who was unaware of the type of treatment of which the patient had received

SECONDARY OUTCOMES:
Nerve conduction study of facial nerve. | 2 months
  Measurment of facial n. coduction

REFERENCES:
- [Derived] Khedr EM, Badry R, Ali AM, Abo El-Fetoh N, El-Hammady DH, Ghandour AM, Abdel-Haleem A. Steroid/Antiviral for the treatment of Bell's palsy: Double blind randomized clinical trial. Restor Neurol Neurosci. 2016 Nov 22;34(6):897-905. doi: 10.3233/RNN-150605. PMID 27689547